CLINICAL TRIAL: NCT01972802
Title: International Cancer of the Head and Neck, Genetics and Environment (InterCHANGE) Study
Acronym: InterCHANGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201006077R
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Evaluate the Association Between Certain Environmental Exposures (e.g. Cigarette Smoking, Alcohol Drinking, Betel Nut Chewing…) and Head and Neck Cancers; Assess the Effect of Genetic Factors, Including Both SNP and Copy Number Variation (CNV) Through Analysis of Both Main Effect and Gene-gene Interaction
Keywords: HEAD AND NECK
MeSH Terms: conditions — Alcohol Drinking; Head and Neck Neoplasms; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BLOOD 20ML, Fresh (biopsy)samples, Oral scrape
Oversight: Data Monitoring Committee: No

SUMMARY:
Our overall objective is to understand the role of lifestyle factors, genetics and HPV infection in the development and prognosis of head and neck cancer particularly in Asia.

ELIGIBILITY:
Inclusion Criteria:

Age 18~80 Incident head and neck cancer patients

* Oral, oropharynx and hypopharynx (C00-C14)
* Laryngreal cancer (C32)
* *Esophageal cancer if possible (C15)

Exclusion Criteria:

* Salivary gland (C07-C08)
* Nasopharynx (C11)
* Thyroid (C79.3)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NTUH HEAD AND NECK PATIENT AND CONTROLS
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
head and neck cancer risk factor | Four years
  evaluate the association between certain environmental exposures (e.g. cigarette smoking, alcohol drinking, betel nut chewing…) and head and neck cancers,assess the effect of genetic factors, including both SNP and copy number variation (CNV) through analysis of both main effect and gene-gene interaction

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jen Lou, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Tiapei, Taipei, Taiwan